CLINICAL TRIAL: NCT05572645
Title: Pyrotinib Plus Trastuzumab Versus Pertuzumab Plus Trastuzumab in HER2-Positive Metastatic Breast Cancer: a Multicenter, Retrospective Study
Brief Title: Pyrotinib Plus Trastuzumab Versus Pertuzumab Plus Trastuzumab
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-21
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Pyrotinib; Trastuzumab; Pertuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Trastuzumab; pertuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PyroH: treatment based on Pyrotinib(320-400 mg, po, qd) Plus Trastuzumab(8 mg/kg q3w, and then 6 mg/kg q3w)
  Interventions: Drug: Pyrotinib Plus Trastuzumab
- PertH: treatment based on Pertuzumab(840mg q3w, and then 420 mg q3w) Plus Trastuzumab(8 mg/kg q3w, and then 6 mg/kg q3w)
  Interventions: Drug: Pertuzumab Plus Trastuzumab

INTERVENTIONS:
Drug: Pyrotinib Plus Trastuzumab — treatment based on Pyrotinib(320-400 mg, po, qd) Plus Trastuzumab(8 mg/kg q3w, and then 6 mg/kg q3w)
  Groups: PyroH
Drug: Pertuzumab Plus Trastuzumab — treatment based on Pertuzumab(840mg q3w, and then 420 mg q3w) Plus Trastuzumab(8 mg/kg q3w, and then 6 mg/kg q3w)
  Groups: PertH

SUMMARY:
Pyrotinib Plus Trastuzumab Versus Pertuzumab Plus Trastuzumab

DETAILED DESCRIPTION:
This is a retrospective study aiming to explore the efficacy and safety of Pyrotinib Plus Trastuzumab Versus Pertuzumab Plus Trastuzumab in patients with HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* HER2+ MBC patients scored +3 by immunohistochemical (IHC) analysis or scored +2 and the result of fluorescence in situ hybridization was positive.
* Patients received Pyrotinib(320-400 mg, po, qd) plus Trastuzumab(8 mg/kg q3w, and then 6 mg/kg q3w) or Pertuzumab(840mg q3w, and then 420 mg q3w) plus Trastuzumab(8 mg/kg q3w, and then 6 mg/kg q3w) for at least one cycle, starting from Jan 2018 to Sep 2022.
* Patients had complete medical records. All data were retrospectively collected from medical records of individual institutions.

Exclusion Criteria:

* Incomplete medical history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Adverse Events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] You S, Xie Y, Sang D, Luo T, Yuan P, Xu F, Wang B. Comparing pyrotinib with trastuzumab and pertuzumab with trastuzumab for HER2-positive metastatic breast cancer: a retrospective, multicenter analysis. Front Endocrinol (Lausanne). 2023 Dec 11;14:1325540. doi: 10.3389/fendo.2023.1325540. eCollection 2023. PMID 38149099